CLINICAL TRIAL: NCT00415571
Title: Efficacy and Safety of Fispemifene in the Treatment of Hypogonadal Men With Erectile Dysfunction Unresponsive to PDE5 Inhibitors: An 8-Week, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Efficacy and Safety Evaluating Fispemifene in the Treatment of Hypogonadal Men With Erectile Dysfunction Unresponsive to PDE5 Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: QuatRx Pharmaceuticals Company (Industry)
Collaborators: Hormos Medical (Industry)
Responsible Party: Janice Margulies/ Development Scientist, QUATRx
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101-50608
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Hypogonadism; Erectile Dysfunction
Keywords: Hypogonadism; Erectile Dysfunction
MeSH Terms: conditions — Hypogonadism; Erectile Dysfunction | interventions — fispemifene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Fispemifene (once daily for 8 weeks)

SUMMARY:
The objective of the study is to assess and compare the preliminary efficacy, safety and tolerability of fispemifene 300 mg and placebo given once daily for 8 weeks in the treatment of hypogonadal men with erectile dysfunction (ED) unresponsive to PDE5 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Hypogonadal (morning total testosterone levels ≤400 ng/dl) men age ≥20 with ED who are unresponsive to PDE5 inhibitors, as demonstrated by International Index of Erectile Function (IIEF) results for 28-day lead in period.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2006-12; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change in the IIEF erectile function domain score from baseline to Week 8/Early Termination;
Change in total testosterone levels from baseline to Week 8/Early Termination

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Radiant Research, Birmingham, Alabama
  - Genova Clinical Research, Tucson, Arizona
  - HealthStar Research, Hot Springs, Arkansas
  - Genesis Research International, Longwood, Florida
  - Renstar Medical Research, Ocala, Florida
  - Radiant Research, West Palm Beach, Florida
  - Regional Urology, Shreveport, Louisiana
  - Office of Stephen Miller, Las Vegas, Nevada
  - Hamilton Urology, Hamilton, New Jersey
  - Center for Urologic Research of WNY, LLC, Williamsville, New York
  - Metrolina Urology Clinic, Charlotte, North Carolina
  - NorthEast Urology research, Concord, North Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Radiant Research, San Antonio, Texas

REFERENCES:
- [Background] Feldman HA, Goldstein I, Hatzichristou DG, Krane RJ, McKinlay JB. Impotence and its medical and psychosocial correlates: results of the Massachusetts Male Aging Study. J Urol. 1994 Jan;151(1):54-61. doi: 10.1016/s0022-5347(17)34871-1. PMID 8254833
- [Background] NIH Consensus Conference. Impotence. NIH Consensus Development Panel on Impotence. JAMA. 1993 Jul 7;270(1):83-90. No abstract available. PMID 8510302
- [Background] Johannes CB, Araujo AB, Feldman HA, Derby CA, Kleinman KP, McKinlay JB. Incidence of erectile dysfunction in men 40 to 69 years old: longitudinal results from the Massachusetts male aging study. J Urol. 2000 Feb;163(2):460-3. PMID 10647654
- [Background] Campbell HE. Clinical monograph for drug formulary review: erectile dysfunction agents. J Manag Care Pharm. 2005 Mar;11(2):151-71. doi: 10.18553/jmcp.2005.11.2.151. PMID 15766322
- [Background] Salonia A, Rigatti P, Montorsi F. Sildenafil in erectile dysfunction: a critical review. Curr Med Res Opin. 2003;19(4):241-62. doi: 10.1185/030079903125001839. PMID 12841917
- [Background] Bhasin S, Cunningham GR, Hayes FJ, Matsumoto AM, Snyder PJ, Swerdloff RS, Montori VM. Testosterone therapy in adult men with androgen deficiency syndromes: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2006 Jun;91(6):1995-2010. doi: 10.1210/jc.2005-2847. Epub 2006 May 23. PMID 16720669
- [Background] Albrecht-Betancourt M, Hijazi RA, Cunningham GR. Androgen replacement in men with hypogonadism and erectile dysfunction. Endocrine. 2004 Mar-Apr;23(2-3):143-8. doi: 10.1385/ENDO:23:2-3:143. PMID 15146093
- [Background] Shabsigh R. Testosterone therapy in erectile dysfunction and hypogonadism. J Sex Med. 2005 Nov;2(6):785-92. doi: 10.1111/j.1743-6109.2005.00139.x. PMID 16422803
- [Background] Kalinchenko SY, Kozlov GI, Gontcharov NP, Katsiya GV. Oral testosterone undecanoate reverses erectile dysfunction associated with diabetes mellitus in patients failing on sildenafil citrate therapy alone. Aging Male. 2003 Jun;6(2):94-9. PMID 12898793
- [Background] Aversa A, Isidori AM, Spera G, Lenzi A, Fabbri A. Androgens improve cavernous vasodilation and response to sildenafil in patients with erectile dysfunction. Clin Endocrinol (Oxf). 2003 May;58(5):632-8. doi: 10.1046/j.1365-2265.2003.01764.x. PMID 12699447
- [Background] Shabsigh R, Kaufman JM, Steidle C, Padma-Nathan H. Randomized study of testosterone gel as adjunctive therapy to sildenafil in hypogonadal men with erectile dysfunction who do not respond to sildenafil alone. J Urol. 2004 Aug;172(2):658-63. doi: 10.1097/01.ju.0000132389.97804.d7. PMID 15247755
- [Background] Yassin AA, Saad F, Diede HE. Testosterone and erectile function in hypogonadal men unresponsive to tadalafil: results from an open-label uncontrolled study. Andrologia. 2006 Apr;38(2):61-8. doi: 10.1111/j.1439-0272.2006.00712.x. PMID 16529577